CLINICAL TRIAL: NCT06393088
Title: Clinical Trial to Establish the Safety and Efficacy of the invisaRED® IR REHAB Device When Used as an Adjunctive Therapy for Nociceptive Musculoskeletal Pain
Brief Title: Clinical Trial of the invisaRED® IR REHAB Device When Used as an Adjunctive Therapy for Nociceptive Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IR Technology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR_REHAB_Clinical_Trial
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Nociceptive Pain; Musculoskeletal Pain
Keywords: Low level laser therapy; photobiomodulation; dual frequency; red; near infrared; light
MeSH Terms: conditions — Nociceptive Pain; Musculoskeletal Pain; Erythema

STUDY DESIGN:
Intervention Model Description: The trial will compare results between two groups; the first will be treated using the invisa-RED Technology IR REHAB and the second group with a sham device. The trial will be conducted employing a single blind study methodology; participants will not know to which trial group they have been assigned. Participants will undergo six (6) therapy sessions each using a standardized 15 minute protocol. At each of the therapy sessions; the participant will be asked to record their pain level before the treatment session and then in the same manner after the treatment using a Visual Analog Scale (VAS). The results from the two groups will be statistically analyzed to determine the efficacy of the invisa-RED Technology IR REHAB as an adjunctive therapy for musculoskeletal pain. Any medical errors will be included in the statistical analysis.
Who Masked: Participant
Masking Description: All individuals participating in the trial will be assigned a participant number. Subsequently all clinical records and reports will reference only the participant number, ensuring that participants remain anonymous.
  Because of the low number of trial participants, only paper records will be maintained for all clinical and personal data. Records will be kept in locked storage and physical access will only be on a need to know basis. A participants' personal data correlating the participating individuals name and the trial participants Identifying Number will only be available to the principal investigator, clinical staff, and the trial administrator. All analytics will be performed on securely encrypted devices using only data masked or redacted of any personal information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IR REHAB Device (Experimental): Participants will receive 6 treatments of 15 minutes each with an active IR REHAB device over the period of three weeks.
  Interventions: Device: IR REHAB
- Sham Device (Sham Comparator): Participants will receive 6 treatments of 15 minutes each with a disabled (sham) IR REHAB device over the period of three weeks.
  Interventions: Device: Sham

INTERVENTIONS:
Device: IR REHAB — Participants undergo therapy sessions with active, dual frequency, low level laser therapy device
  Arms: IR REHAB Device
Device: Sham — Participants undergo therapy sessions with disabled device producing no laser energy
  Arms: Sham Device

SUMMARY:
This is a trial to measure the effectiveness and safety of the invisa-RED® IR REHAB device. The researchers will compare the muscle and joint pain relief of participants who are treated with the real machine, to those treated with a non-working "look-a-like" device. If there is a significant difference of pain relief between those treated with the real machine and those treated with the 'look-a-like' device and no safety issues are discovered, the researchers will be able to assume the IR REHAB device is safe and effective for the treatment of muscle and joint pain.

DETAILED DESCRIPTION:
Clinical Trial to Establish the Safety and Efficacy of the IR REHAB Device When Used as an Adjunctive Therapy for Nociceptive Musculoskeletal Pain

Purpose of the Study

The trial is designed to provide data with which to evaluate the efficacy and safety of the invisa-RED® IR REHAB Low-level Laser Therapy (LLLT) device as compared with a sham device when used for the adjunctive treatment of musculoskeletal pain . This will be a single blind trial of two groups of equal number; one group will be treated as usual, the other treated using a sham device. At the conclusion of the trial; results from the two groups will be statistically analyzed to determine the efficacy of the IR REHAB machine for the adjunctive treatment of musculoskeletal pain .

"Musculoskeletal pain is a challenging condition for both patients and physicians. Many adults have experienced one or more episodes of musculoskeletal pain at some time of their lives, regardless of age, gender, or economic status. It affects approximately 47% of the general population. Of those, about 39-45% have long-lasting problems that require medical consultation. Inadequately managed musculoskeletal pain can adversely affect quality of life and impose significant socioeconomic problems."

Monitoring Plan

The study is classified as a minimal risk trial of short duration therefore a detailed plan for monitoring the data for participant safety is not required.

Data Storage and Security

All individuals participating in the trial will be assigned a participant number. Subsequently all clinical records and reports will reference only the participant number, ensuring that participants remain anonymous.

Because of the low number of trial participants, only paper records will be maintained for all clinical and personal data. Records will be kept in locked storage and physical access will only be on a need to know basis. A participants' personal data correlating the participating individuals name and the trial participants Identifying Number will only be available to the principal investigator, clinical staff, and the trial administrator. All analytics will be performed on securely encrypted devices using only data masked or redacted of any personal information.

Risk/Benefit Assessment

Applying the test for the determination of risk established by the FDA Regulation referred to as the "Common Rule" found in 45 Code of Federal Regulations (CFR) 46, Subpart A the rule states;

"Minimal risk means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests.

The researchers have determined that only a minimal risk is presented to participants of the trial.

All persons interviewed for the trial will be selected using the established invisaRED Technologies IR REHAB guidelines for indications and contraindications. Combining the guidelines for indications and contraindications with the thorough classroom review and "hands on training " for clinicians who will be conducting the trial, the risk is best compared to exposure to sunlight.

Subjects of the study receiving the invisaRED Technologies IR REHAB therapy may receive the following benefits:

1. Open up blood vessels to ease swelling
2. Help the immune system create more chemicals that heal tissue
3. Build more connective tissue in injured area
4. Trigger endorphins, natural hormones that ease pain
5. Drug free therapy without a chance of addiction
6. The therapy is noninvasive
7. There are no known side effects

Subject Identification, Recruitment And Consent/Assent

At roadway intersections in close proximity to the research facility signs will be erected containing the verbiage: "Pain and Injury Study, No Cost, Call 770 988-5594" in order to recruit study volunteers from the community.

The clinic's primary care patients will also be provided an opportunity to volunteer for consideration as a trial participant.

The primary investigator will conduct all subject interviews and obtain informed consent. A thorough disclosure of all clinical process, contraindications, and any risk will be discussed with candidates for the trial.

There shall be no cost incurred by candidates for inclusion in the study or individuals selected to participate in the study.

No monetary remuneration will be offered participants in the study. However a commensurate number of treatments with the "as usual" IR REHAB device will be offered for free to those patients who received treatment using the sham device at the conclusion of the clinical trial. This will provide the participants treated with the sham device the opportunity to undergo therapy using an activated IR REHAB device.

Requirements for Human Subject Protection Training

The Primary Investigator and clinical associates conducting the trial will complete the Collaborative Institutional Training Initiative (CITI) course Good Clinical Practice (GCP) for Clinical Trials with Investigational Drugs and Medical Devices (U.S. FDA Focus).

ELIGIBILITY:
Inclusion Criteria:

The number of participants is projected to be thirty (30).

There will be an equitable distribution of male and female participants.

Women who are pregnant, trying to get pregnant, or nursing will be excluded from the study, as they should not receive Low-level Laser Therapy (LLLT). There is no evidence of harm to a an unborn baby however there have been no safety tests either, so for medical legal reasons we recommend never treating such individuals.

The participants will be 18 years or older.

The ethnicity of the participants will be equitably distributed.

Inclusion criteria will be individuals that may benefit from an adjunctive therapy for musculoskeletal pain.

Exclusion Criteria:

If you are pregnant, trying to get pregnant or nursing laser light therapy should be received only after the end of these conditions. There is no evidence of harm to a an unborn baby however there have been no safety tests either, so for medical legal reasons we recommend never treating areas directly over a developing child.

Individuals with hypertension, light sensitive epilepsy, cancer, heart disease, infectious skin disease, and severe varicose veins should not use this device.

People suffering from infectious and acute disease such as a fever should not use this device.

People who have hemorrhagic disease, vascular ruptures, skin inflammation, or any disease of the skin should not use this device.

Person with a history of lentigines, an autoimmune vascular disease that causes color changes in the legs or arms due to obstruction or stenosis of blood vessels.

A person with a history of erythema, an acquired, long-lasting reticulocyte red and pigmented rash, caused by persistent or repeated exposure to intense heat or infrared radiation.

Persons who are susceptible to or have a history of herpes in the treatment area

Anyone who has experienced problems subsequent to previous laser treatments

People who have immune system dysfunction such as Leukemia, Hemophilia, etc., and light sensitive persons should not use this device.

Use of laser light therapy in the ears, nose, eye, or throat is not recommended.

Individuals with a history of melanoma, raised moles, suspicious lesions, keloid scar formation, or healing problems should not undergo laser light therapy.

Individuals with active infections, open lesions, hives, herpetic lesions, cold sores, or tattoos and permanent make-up in the area of treatment should not undergo laser light therapy.

People who have used isotretinoin (commonly known as Accutane), tetracycline, St. John's Wort, or any photo sensitizing drugs in the last year should not undergo laser light therapy.

Individuals with autoimmune diseases such as Lupus, Scleroderma, or Vitiligo should not undergo laser light therapy.

Individuals who have pacemakers or other electro-stimulation devices surgically implanted should not undergo laser light therapy.

Any insulin dependent individual should consult their physician before undergoing laser light therapy.

All individuals considered "vulnerable" such as children, pregnant women, nursing home residents or other institutionalized persons, students, employees, fetuses, prisoners, and persons with decisional incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajibole Abatunde, MD, Principal Investigator — Midnight Rose LLC dba Abbycare
Locations (1):
- Abbycare Clinic, Woodstock, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Tallawy SN, Nalamasu R, Salem GI, LeQuang JAK, Pergolizzi JV, Christo PJ. Management of Musculoskeletal Pain: An Update with Emphasis on Chronic Musculoskeletal Pain. Pain Ther. 2021 Jun;10(1):181-209. doi: 10.1007/s40122-021-00235-2. Epub 2021 Feb 11. PMID 33575952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Trial recruitment period had a start date of July 22nd and ended on August 7th 2024. (A total of 17 days) All participant recruitment and interviews were conducted at the Abbycare Clinic in Woodstock, GA.
Groups:
- IR REHAB Device: Participants will receive 6 treatments of 15 minutes each with an active IR REHAB device over the period of three weeks.
  IR REHAB: Participants undergo therapy sessions with active, dual wavelength, low level laser therapy device
Period: Overall Study
Arm/Group | IR REHAB Device | Sham Device
Started | 16 | 15
Completed | 16 | 13
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IR REHAB Device | Sham Device | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 7 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 13 | 8 | 21
  Race: Black | 2 | 4 | 6
  Race: Hispanic | 1 | 0 | 1
  Race: Other | 0 | 1 | 1
IR REHAB Clinical Trial Participants [Count of Participants; unit: Participants] | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Measured Change in the Participants Pain Levels
Description: Participants pain levels will be measured using a visual analog scale of 0-100mm where a smaller number indicates a lower perceived pain level and a larger number indicates a higher level of pain. The participant will personally manipulate a visual analog scale with a manual slide indicator to record their pain levels
Time Frame: Participants pain levels will be recorded over a period of three weeks.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | IR REHAB Device | Sham Device
Number analyzed (Participants) | 16 | 13
Score on a scale | 61.46 [47.70 to 72.63] | 19.79 [4.89 to 37.34]
Statistical Analysis 1: Comparison: IR REHAB Device vs Sham Device; Null Hypothesis: There is not a statistically significant difference in nociceptive musculoskeletal pain when using an IR REHAB device when compared with a sham (placebo) device as a therapy in an approved and standardized clinical protocol; Test type: Superiority — It was calculated that 24 participants randomized 1:1 between 2 arms would have at least an 85% power to detect a difference in pain relief of 30 points as measured using a Visual Analog Device. The actual difference in the mean of the change in pain level, as measured using a Visual Analog Scale, between the two independent groups is 41.67. Results of the post trial calculation was a 95.7% power to detect the difference in pain relief using 29 randomized participants; p < 0.01, t-test, 2 sided — The threshold is P-value <.0.05 for statistical significance A bootstrap N=20,000 was used for all estimates; Mean Difference (Net) = 41.67, 95% CI 2-sided [20.15 to 61.67]

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | IR REHAB Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 0/16 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT06393088/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT06393088/ICF_001.pdf